CLINICAL TRIAL: NCT06821659
Title: Safety and Efficacy of Universal CAR-T Cells (UWD-CD19) Combined with Immunosuppressants in the Treatment of Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20250037
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Systemic Lupus Erthematosus; Systemic Sclerosis (SSc); Inflammatory Myopathies; ANCA Associated Vasculitis (AAV); Sjogren Syndrome
MeSH Terms: conditions — Scleroderma, Systemic; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-CD19 CAR-T (UWD-CD19) (Experimental)
  Interventions: Biological: anti-CD19 CAR-T cells

INTERVENTIONS:
Biological: anti-CD19 CAR-T cells — UWD-CD19

SUMMARY:
Autoimmune diseases refer to a common category of diseases caused by the immune system reacting to self-antigens, leading to tissue damage. Autoimmune diseases encompass a wide variety of conditions, such as systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis, inflammatory myopathies, ANCA-associated vasculitis. Current treatments for autoimmune diseases include glucocorticoid, immunosuppressants, and biologics. B cell-driven humoral immune abnormalities are a central pathogenic mechanism in many autoimmune diseases. When autoreactive B cells are excessively activated, they produce large amounts of autoantibodies and immune complexes. These antibodies and immune complexes can cause damage to various tissues and organs, leading to the development of multiple autoimmune diseases. Therefore, targeting B cells to treat autoimmune diseases is an attractive therapeutic strategy. Clinical studies are exploring the use of CD19-targeting CAR-T cells for the treatment of autoimmune diseases, and their therapeutic efficacy has been demonstrated. In this study, we investigate the safety and efficacy of universal CD19-targeting CAR T cells in the treatment of autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years (inclusive), male or female.
2. >40kg.
3. Diagnosed with refractory autoimmune disease, defined as: Ineffectiveness of conventional treatment for more than 6 months, or Disease activity recurrence after remission. Definition of conventional treatment: Use of glucocorticoids and any of the following immunosuppressants or biologics: cyclophosphamide, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, telitacicept, etc.
4. Currently receiving one or more standard therapies at a stable dose, including glucocorticoids, antimalarials, immunosuppressants, or biologics. If the subject is receiving glucocorticoids, the following conditions must be met: During screening and the screening period, the maximum dose of glucocorticoids is 30 mg/day prednisone (or an equivalent dose). The glucocorticoid dose must remain stable for ≥7 days before screening, and during the screening period, the dose adjustment must not exceed >5 mg/day prednisone (or an equivalent dose). If the subject is receiving antimalarials and/or conventional immunosuppressants: The treatment must have started ≥12 weeks before screening. The medication dose must remain stable for ≥8 weeks before screening and throughout the screening period. Before cell infusion, other immunosuppressants (excluding hydroxychloroquine), including belimumab, telitacicept, CD20 monoclonal antibodies, or other biologic immunosuppressants, must be discontinued for at least 5 half-lives.
5. Female participants of childbearing potential and male participants with female partners of childbearing potential must use medically approved contraceptive methods or practice abstinence during the study treatment period and for at least 6 months after the study. Female participants of childbearing potential must have a negative serum HCG test within 7 days before enrollment and must not be breastfeeding.
6. Willing to participate in the trial and sign the informed consent form.

Disease-Specific Inclusion Criteria:

Systemic Lupus Erythematosus (SLE):

1. Meets the 2019 EULAR/ACR classification criteria for SLE.
2. ANA titer ≥1:80, or positive for anti-dsDNA and/or anti-Sm antibodies.
3. Disease activity score (SLEDAI-2000) ≥8.

Sjögren's Syndrome:

1. Meets the 2002 AECG criteria or the 2016 ACR/EULAR classification criteria for primary Sjögren's syndrome.
2. Disease activity score (ESSDAI) ≥5.
3. Positive for anti-SSA/Ro antibodies.

Systemic Sclerosis (SSc):

1. Meets the 2013 EULAR/ACR classification criteria for systemic sclerosis.
2. Classified by Leroy and Medsger as limited or diffuse cutaneous subsets.
3. At screening, mRSS >10; and/or active interstitial lung disease (ILD), defined as: High-resolution computed tomography (HRCT) showing ground-glass opacities. Pulmonary function tests (FVC or DLCO) <70% of predicted values.

Idiopathic Inflammatory Myopathies (IIM):

1. Meets the 2017 EULAR/ACR classification criteria for inflammatory myopathies (including dermatomyositis, polymyositis, antisynthetase syndrome, and necrotizing myopathy).
2. For patients with muscle involvement: a. MMT-8 score <142 and at least two abnormal findings among the following core measures: PhGA or PtGA scores ≥2. Extramuscular disease activity score ≥2. HAQ total score ≥0.25. Muscle enzyme levels ≥1.5 times the upper normal limit. b. Alternatively, MMT-8 ≥142 but with active ILD (HRCT showing ground-glass opacities).
3. Positive for myositis-specific antibodies.

ANCA-Associated Vasculitis (AAV):

1. Meets the 2022 ACR/EULAR diagnostic criteria for ANCA-associated vasculitis, including microscopic polyangiitis, granulomatosis with polyangiitis, or eosinophilic granulomatosis with polyangiitis.
2. Positive for ANCA antibodies (current or historical).
3. Birmingham Vasculitis Activity Score (BVAS) ≥15 (out of 63), indicating active vasculitis.

Exclusion Criteria:

1. Subjects with a history of alcohol abuse or substance abuse within the past 24 weeks;
2. Subjects with other psychiatric disorders such as schizophrenia or major depressive disorder;
3. Subjects with a history of malignancies other than B-cell lymphoma;
4. Subjects with overlapping diseases that affect the assessment of disease activity;
5. Subjects with infections such as human immunodeficiency virus (HIV), hypogammaglobulinemia, T-cell deficiency virus infection, or chronic hepatitis B or C;
6. Subjects with known active tuberculosis (TB) infection or bacterial infections;
7. Subjects with a history of myocardial infarction, cardiac angioplasty or stent placement, unstable angina, active arrhythmia, or other clinically significant heart diseases within 6 months prior to screening;
8. Subjects with a history of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to screening;
9. Subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) levels ≥3×ULN, or bilirubin >1.5×ULN, excluding abnormalities caused by theautoimmune disease;
10. Subjects with chronic kidney failure stage 4 or above, defined as an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² or serum creatinine >2.5 mg/dL;
11. At the screening visit, subjects with any of the following significant hematologic abnormalities caused by bone marrow suppression, excluding abnormalities due to the autoimmune disease:

    1. Hemoglobin <70 g/L;
    2. Absolute neutrophil count <500/mm³;
    3. Platelet count <50,000/mm³;
12. Subjects with a history of severe adverse reactions to cyclophosphamide or fludarabine;
13. Subjects with a prior history of CAR-T therapy;
14. Subjects who received live vaccines within 30 days prior to CAR-T cell infusion;
15. Subjects deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of UWD-CD19 cell injection in the treatment of refractory autoimmune diseases. | 0-6 months
  In this study, adverse events (AEs) are defined as any adverse medical events occurring from the initiation of lymphodepleting chemotherapy to 12 months after the completion of QH103 cell infusion. The incidence, duration, severity, and management of all adverse events occurring after the participants' enrollment will be recorded and evaluated.Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Graft-versus-host disease (GVHD) will be graded based on the criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE, v5.0)
Maximum tolerated dose of UWD-CD19 cells | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2000) score | 90 days, 180 days, 360 days
  The change from baseline in the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2000) score at 90 days, 180 days, 360 days.
Low Lupus Disease Activity State(LLDAS) | 90 days, 180 days, 360 days
  SLE patients who met Low Lupus Disease Activity State(LLDAS)
Systemic Sclerosis Combined Response Index (CRISS) response | 90 days, 180 days, 360 days
  Patients achieve Systemic Sclerosis Combined Response Index (CRISS) response. A responder meets all of the following criteria; otherwise, they are classified as a non-responder. a. Improvement in at least two aspects (≥ 5% increase in ppFVC and/or ≥ 25% decrease in mRSS, HAQ-DI, PtGA, or PhGA); b. Worsening in no more than one aspect (≥ 5% decrease in ppFVC and/or ≥ 25% increase in mRSS, HAQ-DI, PtGA, or PhGA); c. No significant new SSc-related manifestations.
Modified Rodnan Skin Score (mRSS) | 90 days, 180 days, 360 days
  The changes from baseline in the modified Rodnan Skin Score (mRSS).
Vasculitis disease activity assessment (BVAS score) | 90 days, 180 days, 360 days
  The changes from baseline in vasculitis disease activity assessment (BVAS score) for patients with AAV.
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) | 90 days, 180 days, 360 days
  The changes from baseline in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI).
PhGA in patients with inflammatory myopathies | 90 days, 180 days, 360 days
  The changes from baseline in PhGA in patients with inflammatory myopathies
PtGA in patients with inflammatory myopathies | 90 days, 180 days, 360 days
  The changes from baseline in PtGA in patients with inflammatory myopathies
HAQ score in patients with inflammatory myopathies | 90 days, 180 days, 360 days
  The changes from baseline in HAQ score in patients with inflammatory myopathies.
Extramuscular disease activity score | 90 days, 180 days, 360 days
  The change from baseline in Extramuscular disease activity score in patients with inflammatory myopathies
Muscle enzyme levels | 90 days, 180 days, 360 days
  The changes from baseline in muscle enzyme levels in patients with inflammatory myopathies
PK parameters-Cmax | 0-3 months
  Peak concentration (Cmax) in the CAR gene copy number after infusion of QH103
PK parameters-Cmax | 0-3 months
  Peak concentration in CAR-T cell count in peripheral blood
PK parameters-Tmax | 0-3 months
  Time to peak in the CAR gene copy number after infusion of QH103
PK parameters-Tmax | 0-3 months
  Time to peak in CAR-T cell count in peripheral blood after infusion of QH103
PK parameters- AUC0-M3 | 0-3 months
  Area under the concentration-time curve from 0 to 3 months (AUC0-M3) in the CAR gene copy number
PK parameters-AUC0-M3 | 0-3 months
  Area under the concentration-time curve from 0 to 3 months (AUC0-M3) in CAR-T cell count in peripheral blood

IPD SHARING:
Plan to Share IPD: Undecided
This issue has not been decided yet.